CLINICAL TRIAL: NCT01767857
Title: Phase III Double-blinded, Placebo Controlled Study of Xilonix™ for Improving Survival in Metastatic Colorectal Cancer
Brief Title: A Phase III Study of Xilonix in Patients With Advanced Colorectal Cancer
Acronym: XCITE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study crossed the prospective futility boundary of primary endpoint
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-PT023
Record Dates: First submitted 2013-01-08; First posted 2013-01-14 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Pivotal; Colorectal; Survival; Phase 3
MeSH Terms: conditions — Colorectal Neoplasms | interventions — bermekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xilonix (Experimental): MABp1 administered IV every two weeks, plus best supportive care
  Interventions: Drug: Xilonix
- Placebo (Placebo Comparator): Placebo administered IV every two weeks, plus best supportive care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xilonix — Xilonix is a True Human Monoclonal Antibody targeting Interleukin 1 alpha, and is administered intravenously every 2 weeks with best supportive care until clinical or radiographic progression.
  Other Names: MABp1, CA-18C3
  Arms: Xilonix
Drug: Placebo — Placebo plus best supportive care will be administered intravenously every 2 weeks until clinical or radiographic progression.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the True Human Monoclonal antibody Xilonix (MABp1) can prolong the life of colorectal carcinoma patients that are refractory to standard therapy.

DETAILED DESCRIPTION:
In the setting of refractory, metastatic disease a complete resolution of tumor burden is not a reasonable expectation. Instead, the primary goal of anti-tumor therapy at this stage is to eliminate or reduce the symptomatic effects of the tumor, while trying to prolong survival for as long as possible. Due to treatment related morbidity however, few treatment modalities are ideal for this objective. Even with the most recent targeted agents (such as multi-kinase inhibitors), drug related toxicities frequently lead to relatively short treatment durations. With discontinuation of therapy, disease progression is uncontrolled and prognosis is poor.

New agents that control disease progression-while improving tumor-related symptoms, rather than causing significant therapy related morbidity-are vitally needed to treat patients with advanced cancer, including those with colorectal cancer. An approach has been taken to develop such an agent using a monoclonal antibody to block the chronic inflammation involved in both malignant disease progression and constitutional symptoms.

Xilonix™ is expected to inhibit tumor growth and metastasis by interrupting crucial signals that drive angiogenesis and invasiveness. The antibody therapy may also block tumor microenvironment infiltration by leukocytes (such as myeloid suppressor cells) that suppress antitumor immunity, enabling better host immune control of the disease. In addition to local effects on the tumor, Xilonix™ is expected to work systemically to correct the metabolic dysregulation, fatigue and anxiety mediated by chronic inflammatory signaling to the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with pathologically confirmed colorectal carcinoma that is metastatic or unresectable and which is refractory to standard therapy. To be considered refractory, a subject must have experienced progression (or intolerance) after treatment with standard approved regimens including, oxaliplatin, irinotecan flouropyrimidine, bevacizumab, and cetuximab or panitumumab if KRAS wildtype.
2. Subjects will not be treated with any radiation, chemotherapy, or investigational agents while enrolled in this protocol.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0,1, or 2.
4. At least 2 weeks since the last previous cancer treatment including: chemotherapy, radiation therapy, immunotherapy, surgery, hormonal therapy, or targeted biologics.
5. Age ≥ 18 years, male or female subjects.
6. Serum potassium and magnesium levels within institutional normal limits. Total serum calcium or ionized calcium level must be greater than or equal to the lower limit of normal.
7. Adequate renal function, defined by serum creatinine ≤ 1.5 x ULN.
8. Adequate hepatic function
9. Adequate bone marrow function
10. For women of childbearing potential (WOCBP), a negative serum pregnancy test result at Screening.
11. Signed and dated institutional review board (IRB)-approved informed consent before any protocol-specific screening procedures are performed.
12. Patients enrolled must, in the Investigator's judgment, be healthy enough to stay on the clinical trial for three months.

Exclusion Criteria:

1. Mechanical obstruction that would prevent adequate oral nutritional intake.
2. Serious uncontrolled medical disorder, or active infection, that would impair the ability of the patient to receive protocol therapy.
3. Uncontrolled or significant cardiovascular disease, including:
4. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
5. Subjects who have not recovered from the adverse effects of prior therapy at the time of enrollment to ≤ grade 1; excluding alopecia and grade 2 neuropathy.
6. Immunocompromised subjects, including subjects known to be infected with human immunodeficiency virus (HIV).
7. Known hepatitis B surface antigen and/or positive hepatitis C antibody and presence of hepatitis C RNA.
8. History of tuberculosis (latent or active) or positive Interferon-gamma release assay (IGRA).
9. Receipt of a live (attenuated) vaccine within 1 month prior to Screening
10. Subjects with history of hypersensitivity to compounds of similar chemical or biologic composition of XILONIX™.
11. Women who are pregnant or breastfeeding.
12. WOCBP or men whose sexual partners are WOCBP who are unwilling or unable to use an acceptable method of contraception for at least 1 month prior to study entry, for the duration of the study, and for at least 3 months after the last dose of study medication.
13. Weight loss >20% in the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2013-03-31 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (113):
- United States (57):
  - Alabama Oncology, Bruno Cancer Center, Birmingham, Alabama
  - Southern Cancer Center, PC, Mobile, Alabama
  - Northwest Alabama Cancer Center, PC, Muscle Shoals, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - California Cancer Associates for Research and Excellence, Inc. (cCARE), Fresno, California
  - St. Jude Medical Center, Fullerton, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center and LAC USC Medical Center, Los Angeles, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Stanford Cancer Institute, Palo Alto, California
  - American Institute of Research, Whittier, California
  - Advanced Medical Specialists, Miami, Florida
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Swedish Covenant Hospital via Clintell, Inc., Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hines VA Hospital, Hines, Illinois
  - Oncology Specialists, SC, Park Ridge, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Hutchinson Clinic, P.A., Hutchinson, Kansas
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - The Center for Cancer and Blood Disorders, a Division of Regional Cancer Care Associates LLC., Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Park Nicollet, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - North Shore Hematology Oncology Associates, PC, East Setauket, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Weill Cornell Medical College, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - East Carolina Health - Beaufort, Inc. DBA Marion L. Shepard Cancer Center, Washington, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - St. Charles Health System, Inc., Bend, Oregon
  - Good Samaritan Hospital Corvallis - SHOC, Corvallis, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Bon Secours Saint Francis Cancer Center, Greenville, South Carolina
  - Texas Oncology, Bedford, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Dallas, Dallas, Texas
  - Texas Oncology - Grapevine, Grapevine, Texas
  - Millennium Oncology, Houston, Texas
  - Methodist Richardson Cancer Center, Richardson, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Scott & White Healthcare, Temple, Texas
  - Texas Oncology - Longview and Tyler, Tyler, Texas
  - University of TX Health Science Center at Tyler, Tyler, Texas
  - Virginia Oncology Associates, Multiple Locations, Virginia
  - Providence Regional Medical Center Everett, PRCP - Clinical Research, Everett, Washington
  - SCCA - Evergreen Health, Kirkland, Washington
  - University of Washington, Multiple Locations, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - SCCA - Group Health, Seattle, Washington
- Australia (5):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Western Health - Sunshine Hospital, Saint Albans, Victoria
- Austria (4):
  - Hospital Barmherzige Schwestern Linz, Linz
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - LKH Salzburg 3rd Medical Department with Hematology, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, IV. Internal Department, Wels
- Belgium (6):
  - Grand HÃ´pital de Charleroi, Grand Rue 3, Charleroi, Hainaut
  - CHU Dinant Godinne UCL Namur, Yvoir, Namur
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - Domaine Universitaire du Sart Tilman, Liège
- Czechia (4):
  - Masarykův onkologický ústav, Brno
  - Všeobecné fakultní nemocnice v Praze, Onkologická klinika, Prague
  - Thomayerova nemocnice, Onkologická klinika 1.LF TN Praha, Prague
  - Fakultní nemocnice v Motole, Komplexní onkologické centrum, Prague
- Hungary (5):
  - Semmelweis University 1st Dept. Of Internal Medicine, Oncology Division, Budapest
  - "B" Dept. Of Internal Medicine, National Institute of Oncology, Budapest
  - Uzsoki Hospital, Dept. of Oncoradiology, Budapest
  - Dept. Of Oncology, Somogy County Kaposi Mor Teaching Hospital, Kaposvár
  - Dept. Of Oncology, Tolna County Balassa Janos Hospital, Szekszárd
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - FONDAZIONE POLIAMBULANZA â€" ISTITUTO OSPEDALIERO, Brescia
  - A.O. Universitaria Arcispedale S.Anna Di Ferrara, Cona
  - Azienda Ospedaliera University Pisana Uo Oncol Medica 2, Pisa
  - U.O. Oncologia Medica, Pontedera
  - San Giovanni Calibita" Fatebenefratelli Hospital, Rome
- Netherlands (3):
  - Academic Medical Centre Amsterdam, Amsterdam
  - Amphia Hospital, Breda
  - University Medical Center Utrecht Heidelberglaan, Utrecht
- Poland (8):
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej-Curie w Bialymstoku Odzial Onkologii Klinicznej, Bialystok
  - Regionalne Centrum Onkologii Szpitala im. Prof. Franciszka Łukaszczyka, Bydgoszcz
  - Szpital Wojewodzki w Gdyni Sp. Z o.o., Szpital Morski im PCK, Gdynia
  - Przychodnia Lekarska "Komed", Konin
  - NZOZ Vesalius, Krakow
  - Samodzielny Publiczny ZOZ MSZ z Warmińsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie, Klinika Gastroenterologii Onkologicznej, Warsaw
  - NZOZ Magodent sp z.o.o., Warsaw
- Spain (10):
  - Instituto OncolÃ³gico Dr. Rosell., Barcelona
  - Hospital Vall Dhebron Edificio Principal Planta Baja, Barcelona
  - Institut CatalÃ d'Oncologia, Hospital Duran i Reynals, Barcelona
  - Institut CatalÃ d'Oncologia, Barcelona
  - Hospital ClÃ-nica Benidorm, Benidorm
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital 12 De Octubre, Madrid
  - CIOCC, Centro Integral OncolÃ³gico Clara Campal, Madrid
  - Hospital Son LlÃ tzer, Palma
  - Hospital Universitario La Fe, Consultas Externas Oncologia, Valencia
- Switzerland (2):
  - Istituto Oncologico della Svizzera Italiania, Bellinzona
  - Kantonsspital GraubÃnden, Chur
- United Kingdom (2):
  - Christie Hospital, Manchester, Greater Manchester
  - The Royal Marsden Hospital, Sutton, Surrey

REFERENCES:
- [Background] Hong DS, Hui D, Bruera E, Janku F, Naing A, Falchook GS, Piha-Paul S, Wheler JJ, Fu S, Tsimberidou AM, Stecher M, Mohanty P, Simard J, Kurzrock R. MABp1, a first-in-class true human antibody targeting interleukin-1alpha in refractory cancers: an open-label, phase 1 dose-escalation and expansion study. Lancet Oncol. 2014 May;15(6):656-66. doi: 10.1016/S1470-2045(14)70155-X. Epub 2014 Apr 17. PMID 24746841

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 643 participants were screened and enrolled in the study. Out of them, only 611 participants have received the study drug and participated in the study while 32 participants never received any study drug.
Groups:
- Xilonix: Participants received 7.5 milligram per kilogram (mg/kg) Xilonix (MABp1) via intravenous (IV) injection once every 2 weeks until evidence of radiographic or clinical progression along with best supportive care (BSC) (up to 18 months).
- Placebo: Participants received placebo via IV injection once every 2 weeks until evidence of radiographic or clinical progression plus BSC (up to 18 months).
Period: Overall Study
Arm/Group | Xilonix | Placebo
Started | 430 | 213
Treated | 411 | 200
Completed | 0 | 0
Not Completed | 430 | 213
Not completed — Adverse Event | 27 | 7
Not completed — Death | 28 | 13
Not completed — Lack of Efficacy | 299 | 151
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 38 | 18
Not completed — Physician Decision | 17 | 10
Not completed — Protocol Terminated | 1 | 0
Not completed — Randomized But Never Treated | 19 | 13

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were randomized and received at least one infusion of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Xilonix | Placebo | Total
Number analyzed (Participants) | 411 | 200 | 611
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.14) | 61.1 (9.98) | 62.3 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 94 | 253
  Male | 252 | 106 | 358
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 2 | 17
  Black or African American | 20 | 8 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 355 | 186 | 541
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Other | 21 | 4 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 18 | 7 | 25
  Austria | 12 | 3 | 15
  Belgium | 49 | 27 | 76
  Czech Republic | 8 | 3 | 11
  England | 7 | 3 | 10
  Hungary | 8 | 3 | 11
  Israel | 4 | 3 | 7
  Italy | 11 | 7 | 18
  Netherlands | 8 | 4 | 12
  Poland | 30 | 18 | 48
  Spain | 118 | 55 | 173
  Switzerland | 3 | 3 | 6
  USA | 135 | 64 | 199
Age (years) [Count of Participants; unit: Participants]
  < 65 years | 229 | 122 | 351
  Between 65 and 75 years | 141 | 64 | 205
  > 75 years | 41 | 14 | 55
  Missing | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival time was defined as the duration from the date of randomization until death or last follow-up. OS was summarized by Kaplan-Meier method and compared between the treatment groups using un-adjusted log-rank test.
Time Frame: Up to 18 months
Population: The modified intent-to-treat (mITT) population included all participants who were randomized and received at least one infusion of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xilonix | Placebo
Number analyzed (Participants) | 411 | 200
Months | 5.6 [4.9 to 6.2] | 5.4 [4.6 to 6.2]
Statistical Analysis 1: Comparison: Xilonix vs Placebo; Test type: Superiority; p = 0.613, Log Rank

2. Secondary Outcome: Change From Baseline in Lean Body Mass (LBM) Measured by Dual-energy X-ray Absorptiometry (DEXA) Scans
Description: Change from baseline in LBM as measured by Dexa scans was reported. DEXA is an X-ray imaging modality used to determine the mass of one material in the presence of another material, using the knowledge of their unique X-ray attenuation at different energies.
Time Frame: Baseline and Week 8
Population: The per protocol (PP) population was defined as participants that had baseline and follow up values for both the DEXA assessment and the European Organization for Research and Treatment of Cancer (EORTC) questionnaire.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Groups:
- Xilonix: Participants received 7.5 mg/kg Xilonix (MABp1) via IV injection once every 2 weeks until evidence of radiographic or clinical progression along with BSC (up to 18 months).
Arm/Group | Xilonix | Placebo
Number analyzed (Participants) | 202 | 94
kilogram (kg) | 0.51 (0.158) | -0.21 (0.231)
Statistical Analysis 1: Comparison: Xilonix vs Placebo; Test type: Superiority; p = 0.011, ANCOVA

3. Secondary Outcome: Change From Baseline in Symptom Scale and Global Health Status/Quality of Life (QoL) Assessed Through the Cancer-specific European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 questionnaire incorporates nine multi-item scales: 5 functional scales (physical, cognitive, role, emotional, and social); 3 symptom scales (pain, fatigue, and appetite loss) and a Global Health Status/QoL scale. Each item, except Global Health Status, is answered on a four-point scale (1-4): 1-not at all, 2-a little, 3-quite a bit, 4-very much. Response to Global Health Status is measured on a 1 to 7 scale. "1" being very poor and "7" being excellent. Each scale (symptom scale [pain, fatigue, and appetite loss] and Global Health Status/Quality of Life [QoL] scale) was linearly transformed to be in range from 0-100 where a higher score represents good health status, while lower scores indicate poor health status. As planned, the data for symptom scales (pain, fatigue, appetite loss) and a Global Health Status/QoL scale was evaluated and reported.
Time Frame: Baseline and Week 8
Population: The PP population was defined as participants that had baseline and follow up values for both the DEXA assessment and the EORTC questionnaire.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Xilonix | Placebo
Number analyzed (Participants) | 202 | 94
Units on a scale
  Global Health Status/Qol | -6.64 (1.392) | -8.16 (2.041)
  Pain | 8.50 (1.707) | 10.27 (2.503)
  Fatigue | 7.42 (1.516) | 8.82 (2.223)
  Appetite Loss | 9.34 (2.010) | 11.84 (2.947)
Statistical Analysis 1: Comparison: Xilonix vs Placebo; Statistical Analysis for Global Health Status/Qol; Test type: Superiority; p = 0.541, ANCOVA
Statistical Analysis 2: Comparison: Xilonix vs Placebo; Statistical Analysis for Pain; Test type: Superiority; p = 0.560, ANCOVA
Statistical Analysis 3: Comparison: Xilonix vs Placebo; Statistical Analysis for Fatigue; Test type: Superiority; p = 0.603, ANCOVA
Statistical Analysis 4: Comparison: Xilonix vs Placebo; Statistical Analysis for Appetite Loss; Test type: Superiority; p = 0.485, ANCOVA

4. Secondary Outcome: Change From Baseline in Platelet Counts
Description: Change from baseline in platelet counts up to Week 8 was evaluated.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: 1000 cells/cubic millimeter
Arm/Group | Xilonix | Placebo
Number analyzed (Participants) | 202 | 94
1000 cells/cubic millimeter | 5.50 (4.721) | 16.19 (7.082)
Statistical Analysis 1: Comparison: Xilonix vs Placebo; Test type: Superiority; p = 0.210, ANCOVA

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from randomization to tumor progression or death. Progressive Disease defined as increase in tumor burden greater than or equals to (>=) 25 (%) percent relative to nadir (minimum recorded tumor burden) confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented. Participants surviving without disease progression at end of study were censored. PFS was compared by Kaplan-Meier method using log-rank test.
Time Frame: Up to 18 Months
Population: The intent-to-treat (ITT) population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xilonix | Placebo
Number analyzed (Participants) | 430 | 213
Months | 2.1 [2.1 to 2.1] | 2.1 [2.0 to 2.1]
Statistical Analysis 1: Comparison: Xilonix vs Placebo; Test type: Superiority; p = 0.768, Log Rank

6. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: The percentage of OR was estimated by dividing the total number of confirmed complete response (CR) and partial response (PR) by the total number of participants randomized where CR was complete disappearance of all lesions (whether measurable or not, and no new lesions); confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented and PR was decrease in tumor burden >= 50 % relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation.
Time Frame: Up to 18 months
Population: The mITT population included all participants who were randomized and received at least one infusion of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Xilonix | Placebo
Number analyzed (Participants) | 411 | 200
Percentage of Participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With Disease Control
Description: Percentage of participants who achieved disease control was estimated by dividing the total number of confirmed CRs, PRs and stable disease (SD) by the total number of participants randomized where CR was complete disappearance of all lesions (whether measurable or not, and no new lesions); confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented, PR was decrease in tumor burden >= 50% relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation and SD defined as not meeting criteria for CR and PR, in absence of Progressive Disease (increase in tumor burden >= 25 % relative to nadir (minimum recorded tumor burden) confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented).
Time Frame: Up to 18 months
Population: The participants with baseline and follow up radiographic assessments were included in this analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Xilonix | Placebo
Number analyzed (Participants) | 296 | 154
Percentage of Participants | 25 | 27.3

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: Safety analysis included the safety population, defined as enrolled participants who received at least one dose of study drug.
Arm/Group | Xilonix | Placebo
All-Cause Mortality (participants affected / at risk) | 28/411 | 13/200
Serious Adverse Events (participants affected / at risk) | 169/411 | 84/200
Other Adverse Events (participants affected / at risk) | 324/411 | 167/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xilonix (N=411) | Placebo (N=200)
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 9 | 6
Anorectal Stenosis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 7 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 2
Large Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Malignant Bowel Obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Oesophageal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal Stenosis (Gastrointestinal disorders) | 0 | 1
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 6 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Adverse Drug Reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 3 | 2
Chest Pain (General disorders) | 2 | 0
Death (General disorders) | 3 | 1
Disease Progression (General disorders) | 21 | 14
Fatigue (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 8 | 5
Localised Oedema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Oedema Peripheral (General disorders) | 3 | 0
Pain (General disorders) | 5 | 0
Performance Status Decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 6 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 2 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 11 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 2 | 0
Liver Disorder (Hepatobiliary disorders) | 0 | 1
Abdominal Abscess (Infections and infestations) | 2 | 0
Catheter Site Abscess (Infections and infestations) | 0 | 1
Catheter Site Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Kidney Infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2
Pneumonia Staphylococcal (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 3 | 4
Septic Shock (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1
Thrombophlebitis Septic (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0
Viral Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 3 | 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 2
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0
Urinary Tract Stoma Complication (Injury, poisoning and procedural complications) | 0 | 1
Urostomy Complication (Injury, poisoning and procedural complications) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 2
Blood Culture Positive (Investigations) | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 5
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Pelvic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 1
Brain Oedema (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 8 | 1
Haematuria (Renal and urinary disorders) | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 2 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pain Management (Surgical and medical procedures) | 1 | 0
Ureteral Stent Removal (Surgical and medical procedures) | 1 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xilonix (N=411) | Placebo (N=200)
Anaemia (Blood and lymphatic system disorders) | 42 | 20
Sinus Tachycardia (Cardiac disorders) | 11 | 10
Abdominal Pain (Gastrointestinal disorders) | 78 | 41
Constipation (Gastrointestinal disorders) | 51 | 31
Diarrhoea (Gastrointestinal disorders) | 45 | 22
Nausea (Gastrointestinal disorders) | 79 | 46
Vomiting (Gastrointestinal disorders) | 46 | 20
Asthenia (General disorders) | 63 | 35
Fatigue (General disorders) | 109 | 60
Oedema Peripheral (General disorders) | 39 | 23
Pyrexia (General disorders) | 38 | 27
Aspartate Aminotransferase Increased (Investigations) | 23 | 6
Blood Alkaline Phosphatase Increased (Investigations) | 20 | 13
Blood Bilirubin Increased (Investigations) | 25 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 84 | 51
Back Pain (Musculoskeletal and connective tissue disorders) | 44 | 27
Headache (Nervous system disorders) | 21 | 13
Insomnia (Psychiatric disorders) | 16 | 10
Proteinuria (Renal and urinary disorders) | 11 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 | 27
Hypertension (Vascular disorders) | 25 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT01767857/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT01767857/SAP_001.pdf